CLINICAL TRIAL: NCT04192227
Title: Comparison of Two Group Wellness Interventions in Partner Caregivers of Individuals With Traumatic Brain Injury: A Randomized Clinical Trial
Brief Title: Comparison of Two Group Wellness Interventions in TBI Partner Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Rehabilitation Hospital of Indiana (Other)
Responsible Party: Principal Investigator, Denise Krch, Senior Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-1076-19
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Traumatic Brain Injury; Partner Caregiver
Keywords: Spouse; Partner; Caregivers; Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wellness Group 1 (Experimental): Administered by wellness facilitator and co-facilitator.
  Interventions: Behavioral: EnHAncing BehavIors through wellness TreatmentS (HABITS)
- Wellness Group 2 (Active Comparator): Administered by wellness facilitator and co-facilitator.
  Interventions: Behavioral: EnHAncing BehavIors through wellness TreatmentS (HABITS)

INTERVENTIONS:
Behavioral: EnHAncing BehavIors through wellness TreatmentS (HABITS) — Six 75-minute sessions via live video conference wherein participants will receive training in areas of health, wellness and quality of life. Classes will be supplemented with independent homework assignments and discussion on a closed social media forum with peers and facilitators.

SUMMARY:
The purpose of this research study is to compare the effect of two different types of group wellness interventions for partner caregivers of individuals with traumatic brain injury (TBI). The study is designed to evaluate how well these treatments can help TBI partner caregivers improve approach/avoidance behaviors.

DETAILED DESCRIPTION:
A multi-site randomized controlled trial will be conducted to evaluate the effectiveness of two different types of group wellness interventions for partner caregivers of individuals with traumatic brain injury (TBI). 92 participants will be recruited. Participants are randomly assigned to one of two wellness groups. Each group will involve six weekly 75-minute live video conference sessions as well as independent homework assignments that will be discussed in closed social media forums with peers and facilitators. Participants will complete self-report measures (approach and avoidance, anxiety, depression, caregiver appraisal, resilience, self efficacy, social integration, quality of life.) prior to intervention participation, within a week of class 6, and at 3-months post-intervention.. Intervention effectiveness will be determined by improvements between baseline and follow-up on a self-report measure of approach/avoidance behaviors.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age.
* read and speak English fluently.
* have been in an intimate relationship with a person with TBI for at least one year prior to their injury.
* partner was discharged from inpatient rehabilitation at least 3 months ago.
* provide care to partner on a daily basis.
* have access to the internet in a private location.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change on Behavioral Inhibition Scale (BIS) | 6 weeks (between pre- and post testing)
  The BIS measures avoidance of aversive stimuli (e.g., anxiety, fear worry)
Change on Behavioral Activation Scale (BAS) | 6 weeks (between pre- and post testing)
  The BAS measures responsiveness to goals, fun, and rewarding stimuli.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rehabilitation Hospital of Indiana, Indianapolis, Indiana
  - Kessler Foundation, East Hanover, New Jersey

IPD SHARING:
Plan to Share IPD: No